CLINICAL TRIAL: NCT03900611
Title: To Investigate the Effects of Peripheral Electrical Stimulation on Cortical Imagining, Electrophysiology and Clinical Profile in Patients With Migraine
Brief Title: Peripheral Electrical Stimulation for Migraine Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-01-001C
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active stimulation (Experimental)
  Interventions: Device: peripheral electrical stimulation
- Sham stimulation (Sham Comparator)
  Interventions: Device: peripheral electrical stimulation
- healthy control (No Intervention)

INTERVENTIONS:
Device: peripheral electrical stimulation — The subjects will undergo 8-week home-based peripheral electrical simulation on the median nerve. The peripheral electrical simulation will be performed once a day for 30 minutes. The stimulation will be active or sham depend on the group assignment.
  Arms: Active stimulation; Sham stimulation

SUMMARY:
Migraine is a common and disabling disease that affects more than 10% of the population worldwide. The prevalence of migraine in Taiwan is around 9.1%. The migraineurs missed 2 workdays due to migraine per year, that is 3.7 million estimated missed workdays in total and an estimated cost of 4.6 billion New Taiwan dollars. In addition, some migraineurs have poor response to the medications or suffer from adverse effects, and may further develop medication-overuse headache. Therefore, in recent years, efforts have been made to develop non-medication treatments, and the number of studies using neuromodulation as an intervention has increased dramatically. Among them, peripheral electrical stimulation has long been a routine treatment for pain in the clinic, and research has also shown its good evidence. In addition, recent studies have shown that peripheral electrical stimulation can also alter the cortical activities. Compared with the proximal brain stimulation, the remote electrical stimulation is safer, more convenient, less expensive and suitable for home use. To date, only one research had focused on the immediate anesthetic effect of remote electrical stimulation whereas the research for migraine prevention is still absent. Therefore, we expect to utilize a more remote electrical stimulation than trigeminal nerve electrical stimulation, which is the commonly used research method nowadays, as an interventional model. In three years, we will recruit 80 migraineurs along with 40 healthy controls and investigate the effects of 8-week home-based remote electrical stimulation on the prevention of migraine and the mechanisms using brain imaging, electrophysiological and biochemical examinations. We also aim to identify the predictors of the responders to remote electrical stimulation. If the effects of remote electrical stimulation are confirmed, as a non-drug neuromodulation management with features of non-invasive, low adverse effects and high accessibility, it will greatly lower the cost of social health care and better improve the quality of life and clinical status of the migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* Migraine:

  1. Diagnosed as migraine by International Classification of Headache Disorder (ICHD-III) criteria
  2. onset before 50 years old
  3. 20-65 yrs.
  4. 4 or more migraine days per month in average
* Healthy control:

  1. devoid of any systemic or neurological diseases

Exclusion Criteria:

1. history of major systemic illness, including uncontrolled hypertension, diabetes, chronic renal insufficiency, autoimmune diseases or malignancies
2. history of neurological disorders which might affect sensation such as previous stroke or peripheral neuropathy
3. pregnancy or lactation
4. epilepsy
5. moderate depressed (BDI>20)
6. using prophylactics for migraine
7. other remote electrical stimulation contraindications, such as open wound, sensory impairment, metal implant
8. other transcranial magnetic stimulation contraindications, such as, high intracranial pressure, cochlear implant, cranial metal implant
9. other magnetic resonance imaging contraindications, such as, pacemaker, stent, metal implant, claustrophobia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
change in migraine or headache days of a month in average | 2 months
  change in migraine or headache days of a month in average
responder rate | 2 months
  responder rate (50% pain reduction from baseline)

SECONDARY OUTCOMES:
change in moderate to severe headache days of a month in average | 2 months
acute headache medication use | 2 months
Beck Depression Inventory | 2 months
modified Migraine Disability Scale | 2 months
  This modified Migraine Disability Scale assesses the migraine related disability in the past 1 month. The total score will be compared and the lower score stands for better outcome.
Patient/Clinical Global Impression of Change | 2 months
  Patient/Clinical Global Impression of Change (PGIC/CGIC) are 7-point scales to assess the improvement by patients themselves and by their clinicians.
Sensory threshold change after treatment | 2 months
  Using quantitative sensory testing (QST) to evaluate the sensory threshold before and after treatment
EEG change after treatment (1) Linear analysis of EEG before and after treatment | 2 months
  power spectal density change of EEG before and after treatment
EEG change after treatment (2) Nonlinear analysis of EEG before and after treatment | 2 months
  functional connectivity change of EEG before and after treatment
fMRI change after treatment | 2 months
  functional connectivity change of fMRI before and after treatment
MRI change after treatment | 2 months
  VBM changes of MRI before and after treatment

IPD SHARING:
Plan to Share IPD: Undecided